CLINICAL TRIAL: NCT02689531
Title: Prospective Observational Study of the Risk Factors for Hospital-Acquired and Ventilator-Associated Bacterial Pneumonia (HABP/VABP)
Brief Title: CTTI Risk Factors for HABP/VABP Study
Acronym: PROPHETIC
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Clinical Trials Transformation Initiative (Other); Food and Drug Administration (FDA) (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00068313
Record Dates: First submitted 2016-02-11; First posted 2016-02-24 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2019-10

CONDITIONS: Pneumonia, Ventilator-Associated; Pneumonia, Bacterial; Pneumonia, Hospital-Acquired
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia, Bacterial; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- High-Risk (Adult =>18 years old): Treated with one or more of the following respiratory modalities for at least 12 continuous hours, either currently or within the prior 7 days:
  * Invasive mechanical ventilation
  * Noninvasive ventilation (BiPAP or CPAP for any indication other than obstructive sleep apnea)
  * High-flow, supplemental oxygen therapy via nasal cannula. Only include systems that using an air/oxygen blender capable of delivering a precise FiO2 level, not just a flow in LPM.
  * High flow supplemental oxygen therapy delivering at least 50% FiO2 via aerosol facemask or tracheostomy collar (mask). Only include systems using an air/oxygen blender capable of delivering a precise FiO2 level, not just a flow in LPM.
  * Supplemental oxygen therapy delivered via either partial or non-rebreather face mask
- Other-ICU/Standard Risk: Patients do not fulfill high-risk criteria, but, are receiving an antibiotic for treatment of lower respiratory tract infection or undifferentiated sepsis.
- High-Risk (Pediatric ≥120 days old and <18 years old): Currently treated with one or more of the following respiratory modalities for at least 24 hours:
  * Invasive mechanical ventilation via endotracheal intubation
  * New initiation of mechanical ventilation, BiPAP or CPAP via tracheostomy
  * Noninvasive ventilation (BiPAP or CPAP for any indication other than obstructive sleep apnea)
  * High-flow, supplemental oxygen therapy delivering at least 1.5LMP with 100% FiO2 via nasal cannula when delivered using an air/oxygen blender capable of delivering a precise FiO2 level, not just a flow in LPM
  * High flow supplemental oxygen therapy delivering at least 50% FiO2 via aerosol facemask or tracheostomy collar (mask) when delivered using an air/oxygen blender capable of delivering a precise FiO2 level, not just a flow in LPM
  * Supplemental oxygen therapy delivered via either partial or non-rebreather face mask
- High-Risk (Pediatric <120 days old): Currently treated with mechanical ventilation via endotracheal intubation for at least 5 days

SUMMARY:
The purpose of this study is to better define the intensive care unit population at highest risk for developing Hospital-Acquired and Ventilator-Associated Bacterial Pneumonia (HABP/VABP).

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study of adult patients (≥18 years old) admitted to ICUs. Generally, all patients admitted to the ICU for any indication will be considered at risk for developing HABP/VABP. A subset of the at-risk patients treated with select respiratory modalities for at least 12 hours will be considered high risk for the development of HABP/VABP, will have baseline data collected, and will be screened daily for antibiotic treatment for suspected pneumonia. Patients not meeting high-risk criteria, "other-ICU patients", will be screened twice weekly for antibiotic treatment for suspected pneumonia.

Once a high-risk subject or other-ICU patient is treated with antibiotics for either a lower respiratory tract infection (LRTI) or undifferentiated sepsis, additional clinical information will be recorded from the subject's medical record. All subjects treated with antibiotics for either indication will subsequently be screened for the development of pneumonia, as defined by the FDA draft guidance document for drug development in HABP/VABP. Subjects who meet the FDA draft guidance definition of pneumonia will have vitals and physiologic data collected and will be followed for 4 days after pneumonia is diagnosed to capture the results of any microbiologic testing and changes to initial antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria (Adult arm => 18 years old):

* Admission to participating ICU
* Hospitalized for >48 hours or admitted <7 days after discharge from an inpatient acute or chronic care facility

High-Risk Inclusion (Adult arm => 18 years old):

Treated with one or more of the following respiratory modalities for at least 12 hours, either currently or within the prior 7 days:

* Invasive mechanical ventilation
* Noninvasive ventilation (BiPAP or CPAP for any indication other than obstructive sleep apnea)
* High-flow, supplemental oxygen therapy via nasal cannula. Only include systems that using an air/oxygen blender capable of delivering a precise FiO2 level, not just a flow in LPM.
* High flow supplemental oxygen therapy delivering at least 50% FiO2 via aerosol facemask or tracheostomy collar (mask). Only include systems using an air/oxygen blender capable of delivering a precise FiO2 level, not just a flow in LPM.
* Supplemental oxygen therapy delivered via either partial or non-rebreather face mask

Other-ICU Inclusion(Adult arm => 18 years old):

All patients who meet ICU and time-frame eligibility criteria, but do not fulfill high-risk criteria, and are receiving an antibiotic for treatment of LRTI or undifferentiated sepsis.

Exclusion Criteria(Adult arm => 18 years old):

* Age <18 years old
* Pregnancy (current) or breastfeeding
* Lung cancer or another malignancy metastatic to the lungs (currently receiving treatment)
* Patient previously enrolled and treated for suspected HABP or VABP (More than CRF Part 1 was previously completed)
* Patient is on comfort measures (e.g. would not receive antibiotics)

Inclusion Criteria (Pediatric Arm: < 18 years old)

* < 18 years old
* Admission to participating ICU or intermediate care unit
* Hospitalized for >48 hours or admitted <7 days after discharge from an inpatient acute or chronic care facility Note: Children and infants with pulmonary and cardiac anomalies are eligible to participate.

High-Risk Inclusion (Pediatric Arm: < 18 years old)

Subjects ≥120 days old and <18 years old:

Currently treated with one or more of the following respiratory modalities for at least 24 hours:

* Invasive mechanical ventilation via endotracheal intubation
* New initiation of mechanical ventilation, BiPAP or CPAP via tracheostomy
* Noninvasive ventilation (BiPAP or CPAP for any indication other than obstructive sleep apnea)
* High-flow, supplemental oxygen therapy delivering at least 1.5LMP with 100% FiO2 via nasal cannula when delivered using an air/oxygen blender capable of delivering a precise FiO2 level, not just a flow in LPM
* High flow supplemental oxygen therapy delivering at least 50% FiO2 via aerosol facemask or tracheostomy collar (mask) when delivered using an air/oxygen blender capable of delivering a precise FiO2 level, not just a flow in LPM
* Supplemental oxygen therapy delivered via either partial or non-rebreather face mask

Subjects <120 days old:

Currently treated with mechanical ventilation via endotracheal intubation for at least 5 days

Standard-Risk Inclusion (Pediatric Arm: < 18 years old) All patients who meet pediatric eligibility criteria, but do not fulfill high-risk criteria, and are receiving an antibiotic for treatment of LRTI or undifferentiated sepsis.

Exclusion Criteria (Pediatric Arm: < 18 years old)

* Known pregnancy (current) or breastfeeding
* Lung cancer or another malignancy metastatic to the lungs (currently receiving treatment)
* Patient previously enrolled and treated for suspected HABP or VABP (More than Pediatric CRF Part 1 was previously completed)
* Patient is on comfort measures (e.g. would not receive antibiotics)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All ICU patients at participating sites hospitalized for >48 hours or admitted <7 days after discharge from an inpatient acute or chronic care facility
Sampling Method: Non-Probability Sample
Enrollment: 7530 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Development of HABP/VABP | Through completion of the study, up to 12 months
  Estimate the rate of HABP/VABP diagnosis in ICU subjects who meet the predetermined high-risk criteria.
Eligibility for typical antibacterial clinical trial | Through completion of the study, up to 12 months
  Estimate the proportion of ICU subjects diagnosed with HABP/VABP who would be eligible for enrollment in a clinical trial of antibacterial therapy for HABP/VABP per FDA draft guidance on HABP/VABP

SECONDARY OUTCOMES:
In enrolled subjects, what factors are associated with the development of hospital acquired or ventilator associated pneumonia. | Through completion of the study, up to 12 months
  Assess the risk factors, comorbid medical illnesses, and treatment exposures associated with the development of HABP/VABP in ICU subjects at high-risk for developing pneumonia using a logistic regression model with age, sex, height (cm), weight (kg), ICU type, admission source, hospital length of stay at the time of screening (calendar days), ICU length of stay at the time of screening, ICU admission diagnosis, aspiration risk, medical history, type and duration of ventilation, enteral nutrition, medications, and other therapies of interest as factors

CONTACTS AND LOCATIONS:
Overall Officials: Vance G Fowler, MD, MHS, Principal Investigator — Duke University
Locations (15):
- United States (15):
  - Birmingham, Alabama
  - Los Angeles, California
  - Chicago, Illinois
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Royal Oak, Michigan
  - St Louis, Missouri
  - Rochester, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Following completion of the study, the results of this research will be written up in a manuscript to be submitted to a scientific journal. The IPD and analysis dataset are available on Vivli.org.
Supporting Information: Study Protocol
Time Frame: The IPD and analysis dataset are available on Vivli.org
Access Criteria: Complete data request process at vivli.org.
URL: https://doi.org/10.25934/PR00008648

REFERENCES:
- [Result] Bergin SP, Coles A, Calvert SB, Farley J, Powers JH, Zervos MJ, Sims M, Kollef MH, Durkin MJ, Kabchi BA, Donnelly HK, Bardossy AC, Greenshields C, Rubin D, Sun JL, Chiswell K, Santiago J, Gu P, Tenaerts P, Fowler VG Jr, Holland TL. PROPHETIC: Prospective Identification of Pneumonia in Hospitalized Patients in the ICU. Chest. 2020 Dec;158(6):2370-2380. doi: 10.1016/j.chest.2020.06.034. Epub 2020 Jun 29. PMID 32615191
- [Result] Bergin SP, Calvert SB, Farley J, Sun JL, Chiswell K, Dieperink W, Kluytmans J, Lopez-Delgado JC, Leon-Lopez R, Zervos MJ, Kollef MH, Sims M, Kabchi BA, Rubin D, Santiago J, Natarajan M, Tenaerts P, Fowler VG, Holland TL, Bonten MJ, Hullegie SJ. PROPHETIC EU: Prospective Identification of Pneumonia in Hospitalized Patients in the Intensive Care Unit in European and United States Cohorts. Open Forum Infect Dis. 2022 May 9;9(7):ofac231. doi: 10.1093/ofid/ofac231. eCollection 2022 Jul. PMID 35836748
- [Result] Ericson JE, McGuire J, Michaels MG, Schwarz A, Frenck R, Deville JG, Agarwal S, Bressler AM, Gao J, Spears T, Benjamin DK Jr, Smith PB, Bradley JS; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee and the Clinical Trials Transformation Initiative. Hospital-acquired Pneumonia and Ventilator-associated Pneumonia in Children: A Prospective Natural History and Case-Control Study. Pediatr Infect Dis J. 2020 Aug;39(8):658-664. doi: 10.1097/INF.0000000000002642. PMID 32150005
- Available data/document: Individual Participant Data Set: VIV00008648 — https://doi.org/10.25934/PR00008648

DOCUMENTS (1):
  • Study Protocol (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT02689531/Prot_000.pdf